CLINICAL TRIAL: NCT05161234
Title: A Clinical Utility Study of PrismRA Testing Therapeutic Response for Rheumatoid Arthritis (DRIVE)
Brief Title: A Clinical Utility Study of PrismRA for Rheumatoid Arthritis
Acronym: DRIVE
Status: Completed | Type: Observational
Sponsor: Scipher Medicine (Industry)
Responsible Party: Sponsor
Other Study IDs: Scipher-RA-005
Record Dates: First submitted 2021-12-03; First posted 2021-12-17 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood will be collected using PrismRA kit consisting of 1 serum separator and 2 PaxGene tubes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A clinical utility study for PrismRA testing therapeutic response in patients with rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 at time of consent
* Patient must meet the criteria for RA as defined by the 2010 ACR/EULAR classification at Visit 1
* Patient has active, moderate to high, RA with a CDAI of >10 at Visit 1
* Patient has swollen and tender joint count of ≥ 2 each, as determined by CDAI assessment at Visit 1 using a 28-joint count
* Patient may participate in additional observational studies concurrently
* Patient is willing and able to complete the informed consent process and comply with study procedures and visit schedule

Exclusion Criteria:

* Patients who are unable to understand the protocol and unable to provide informed consent
* Patients who are not indicated for PrismRA
* Patients who are receiving concurrent treatment with an investigational therapy or have used an investigational therapy less than 4 weeks prior to Visit 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with RA who will have a PrismRA test completed as part of the trial.
Sampling Method: Non-Probability Sample
Enrollment: 613 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2023-12-06 (Actual); Study Completion 2023-12-06 (Actual)

PRIMARY OUTCOMES:
Therapeutic Response | 12-or 24-weeks
  Proportion of moderate to severe disease activity patients that achieve measurable clinical outcomes therapeutic response after initiation of a non-csDMARD therapy

CONTACTS AND LOCATIONS:
Locations (30):
- United States (30):
  - Arizona Arthritis, Chandler, Arizona
  - Medvin Clinical Research//Covina Arthritis Clinic, Covina, California
  - Southland Arthritis, Hemet, California
  - ACRC Studies, Poway, California
  - Medvin Clinical Research//Cohen Medical Center, Thousand Oaks, California
  - Medvin Clinical Research//Foothill Arthritis Clinic, Tujunga, California
  - Medvin Clinical Research/Charles Weidmann, Inc., Van Nuys, California
  - Medvin Clinical Research//Amicus Arthritis, Whittier, California
  - Center for Rheumatology Research, Woodland Hills, California
  - HARAC Research Corp., Avon Park, Florida
  - GNP Research//Mark Jaffe, MD PA, Hollywood, Florida
  - Advanced Clinical Research of Orlando, Ocoee, Florida
  - Rheumatology Associates, PLLC, Louisville, Kentucky
  - Arthritis & Diabetes Clinic, Inc., Monroe, Louisiana
  - Annapolis Rheumatology, Annapolis, Maryland
  - Mid-Atlantic Rheumatology, Glen Burnie, Maryland
  - Advanced Rheumatology, Lansing, Michigan
  - St. Paul Rheumatology, Eagan, Minnesota
  - Innovative Health Research, Las Vegas, Nevada
  - Arthritis and Osteoporosis Consultants of the Carolinas, Charlotte, North Carolina
  - Cape Fear Arthritis Care, Leland, North Carolina
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - Low Country Rheumatology, Summerville, South Carolina
  - Wajeeha Yousaf, MD, PA, Bellaire, Texas
  - Adriana Pop Moody MD Clinic PA// Corpus Christi Rheumatology Clinic, Corpus Christi, Texas
  - Laila Hassan, MD, PA, Houston, Texas
  - Houston Rheumatology & Arthritis Specialists, PLLC, Katy, Texas
  - Main Rheumatology Associates of South Texas, San Antonio, Texas
  - Advanced Rheumatology of Houston, The Woodlands, Texas

DOCUMENTS (2):
  • Study Protocol (2022-10-20): https://cdn.clinicaltrials.gov/large-docs/34/NCT05161234/Prot_002.pdf
  • Statistical Analysis Plan (2022-11-11): https://cdn.clinicaltrials.gov/large-docs/34/NCT05161234/SAP_003.pdf